CLINICAL TRIAL: NCT05488561
Title: Clinical and Molecular Evaluation of Childern With Familial Meditterranean Fever and Their Siblings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nahla Abdelziz Fawy, resident doctor at pediatric department at faculty of medicine sohag university hospital, Sohag University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Soh_Med_22_07_20
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Familial Mediterranean Fever
MeSH Terms: conditions — Familial Mediterranean Fever | interventions — Blood Cell Count; Kidney Function Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CBC with differential ,ESR ,CRP, Amyloid level , FMF gene — leucocytosis , high ESR and CRP ,amyloid level indicates inflammation positive FMF gene indicates having the disease .
  Other Names: liver and kidney function tests

SUMMARY:
Familial Mediterranean fever (FMF ,recurrent polyserositis ,periodic disease) is an autosomal recessive auto inflammatory disease which primarily affect population surrounding the Mediterranean basin (Arabs , Turks ,Armenians, Jews ).Despite its striking symptoms pattern FMF was first described as distinct entity only in 1945.

It is characterized by recurrent attacks of fever , peritonitis ,pleurisy , arthritis , or erysipelas like skin disease. The most dangerous complication of this disease is secondary amyloidosis . FMF diagnosis is mainly clinical, and the genetic testing is indicated to support it . Uncommonly, amyloidosis may develop in individuals carrying two Familial Mediterranean fever gene (MEFV ) mutations without overt clinical symptoms of FMF, a condition designated as phenotype II. Furthermore, two MEFV mutations may be harbored without signs or symptoms of FMF nor of reactive amyloidosis. This 'silent' homozygous or compound heterozygote state is termed phenotype III.

ELIGIBILITY:
Inclusion Criteria:

A- all children diagnosed as FMF according to Tel hashomer criteria aged below 18 years:

The presence of at least 2 of the following 5 criteria after exclusion of other causes can diagnose FMF with high sensitivity:

1. Fever axillary temperature of >38ᵒC, 6-72 h of duration, ≥3 attacks
2. Abdominal pain 6-72 h of duration ≥3 attacks
3. Chest pain 6-72 h duration≥ 3 attacks
4. Arthritis 6-72 h duration ≥3 attacks, oligoarthritis
5. Family history of FMF*(11) B-sisters and brothers of a child with FMF with clinical or subclinical manifestation of FMF.

Exclusion Criteria:

1. Children with other auto inflammatory diseases, or with other diseases.
2. Persons above 18 years old.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
CBC | 12 month
  leucocytosis
amyloid level | 12 month
  high in untreated patients
FMF gene | 12 month
  positive or negative

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alghamdi M. Familial Mediterranean fever, review of the literature. Clin Rheumatol. 2017 Aug;36(8):1707-1713. doi: 10.1007/s10067-017-3715-5. Epub 2017 Jun 18. PMID 28624931
- [Background] Cakan M, Karadag SG, Tanatar A, Sonmez HE, Ayaz NA. The Value of Serum Amyloid A Levels in Familial Mediterranean Fever to Identify Occult Inflammation During Asymptomatic Periods. J Clin Rheumatol. 2021 Jan 1;27(1):1-4. doi: 10.1097/RHU.0000000000001134. PMID 31524848
- [Background] Ozdogan H, Ugurlu S. Familial Mediterranean Fever. Presse Med. 2019 Feb;48(1 Pt 2):e61-e76. doi: 10.1016/j.lpm.2018.08.014. Epub 2019 Jan 25. PMID 30686512
- [Background] Talaat HS, Sheba MF, Mohammed RH, Gomaa MA, Rifaei NE, Ibrahim MFM. Genotype Mutations in Egyptian Children with Familial Mediterranean Fever: Clinical Profile, and Response to Colchicine. Mediterr J Rheumatol. 2020 Jun 15;31(2):206-213. doi: 10.31138/mjr.31.2.206. eCollection 2020 Jun. PMID 32676558